CLINICAL TRIAL: NCT05097443
Title: A Multi-center and Prospective Clinical Study of Orelabrutinib, Rituximab and Combination Chemotherapy in Patients With Newly-diagnosed Aggressive B-cell Non-Hodgkin Lymphoma
Brief Title: Orelabrutinib, Rituximab and Combination Chemotherapy in Newly-diagnosed Aggressive B-cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Department of Hematology, Shandong Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-NHL001
Record Dates: First submitted 2021-10-26; First posted 2021-10-28 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; High Grade B-Cell Lymphoma, Not Otherwise Specified; Diffuse Large B-cell Lymphoma; Mantle Cell Lymphoma; B-cell NonHodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib+R+chemotherapy (Experimental): Orelabrutinib+R-CHOP;Orelabrutinib+R-DA-EPOCH;Orelabrutinib+R-HD MTX；Orelabrutinib+R+other regimens
  Interventions: Drug: Orelabrutinib+R-CHOP; Orelabrutinib+R-DA-EPOCH; Orelabrutinib+R-HD MTX;Orelabrutinib+R+other chemotherapies

INTERVENTIONS:
Drug: Orelabrutinib+R-CHOP; Orelabrutinib+R-DA-EPOCH; Orelabrutinib+R-HD MTX;Orelabrutinib+R+other chemotherapies — Orelabrutinib+R-CHOP： Orelabrutinib 150mg qd; R-CHOP：Rituximab 375mg/m2 d0, Cyclophosphamide 750mg /m2 d1, Doxorubicin 50mg /m2 or Doxorubicin liposome 30-40 mg /m2 d1, Vincristine 1.4mg /m2 or Vindesine 3mg /m2 d1, Prednisone 100mg d1-5.
  Orelabrutinib+R-DA-EPOCH： Orelabrutinib 150mg qd； R-DA-EPOCH：Rituximab 375mg/m2 d0, Etoposide 50mg/ m2, Epirubicin 15mg/ m2, Vincristine 0.4mg/ m2, d1-4, Cyclophosphamide 750mg/ m2 d5, Prednisone 60mg/ m2 d1-5.
  Orelabrutinib+R-HD-MTX: Orelabrutinib 150mg qd; R-HD-MTX: Rituximab 375mg/m2 d0, Methotrexate 3.5g/ｍ2 d1.
  Orelabrutinib+ R+other regimens: Orelabrutinib 150mg qd； R+other regimens: Rituximab 375mg/m2 d0. The dose of other drugs depends on the regimen.
  All regimens follow every 21 days is one cycle, which can be extended to 28 days per cycle according to patients' specific tolerance.
  Dose adjustments of Orelabrutinib are allowed. The initial dose is 150 mg, QD, while the first adjustment is 100 mg, QD and the second adjustment is 50 mg, QD.

SUMMARY:
B-cell non-Hodgkin's lymphoma (B-NHL) is the most common type of NHL. Although novel immunotherapies represented by anti-CD20 monoclonal antibodies and CAR-T cell therapies have significantly improved the prognosis of B-NHL patients, there are still nearly one-third of patients who are resistant to initial treatment or relapse after remission. R-CHOP combined with novel drugs was expected to improve the prognosis. Therefore, this study aimed to investigate the potential of Orelabrutinib combined with Rituximab and chemotherapy.

DETAILED DESCRIPTION:
Non-Hodgkin lymphoma (NHL), with high aggressiveness and mortality, is one of the top ten high-incidence tumors in the world and is among the ten most prevalent cancers worldwide with the fastest growing incidence. B-cell non-Hodgkin's lymphoma (B-NHL) is the most common type of NHL. Although novel immunotherapies represented by anti-CD20 monoclonal antibodies and CAR-T cell therapies have significantly improved the prognosis of B-NHL patients, there are still nearly one-third of patients who are resistant to initial treatment or relapse after remission. In recent years, the continuous emergence of various novel targeted agents has provided new hope for the treatment of B-NHL.

Brutons tyrosine kinase (BTK) is a vital protein for immune B cell function, and a core switch of B cell growth, controlling cellular proliferation, differentiation, apoptosis and migration. BTK inhibitors were available as a breakthrough therapy at the end of 2013, providing a possibility of cure in patients with B-NHL. Orelabrutinib is a highly selective novel BTK inhibitor, and its latest clinical data was announced at the 62nd Annual Meeting of the American Society of Hematology (ASH) on Dec 7, 2020. In two clinical studies targeting relapsed/refractory mantle cell lymphoma (MCL) and relapsed/refractory chronic lymphocytic leukemia (CLL)/small cell leukemia (SLL), orelabrutinib showed a favorable overall remission rate (ORR) and safety. In a phase II clinical study on the treatment of relapsed/refractory CLL/SLL, at a median follow-up of 14.3 months, ORR was 91.3%. The median time to response was 1.87 months, and the median PFS or DOR was not reached. In a phase II clinical study on the treatment of relapsed/refractory MCL, at a median follow-up of 16.4 months, ORR was 87.9%. 93.9% of patients achieved disease control. However, the efficacy of orelabrutinib in highly aggressive B-cell lymphoma remains to be further studied.

Therefore, we present this study protocol to add orelabrutinib to the first-line treatment of highly aggressive B-NHL, applying orelabrutinib+R-CHOP/R-EPOCH/R-HD-MTX/R-other regimens, to clarify the efficacy of orelabrutinib+R-CHOP/R-EPOCH/R-HD-MTX/R-other regimens and explore a set of potent and safe treatments for B-NHL patients with high risks and further improve the prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, gender not limited
2. Newly and histologically diagnosed aggressive B-NHL
3. Patients who have not received systematic chemotherapy or immunotherapy;
4. Patients with at least ≥1 tumor foci with a measurable maximum axis exceeding 1.5 cm;
5. Eastern cancer collaboration group(ECOG) physical status score: 0-2
6. Major organ functions meet the following criteria:

   1. Blood routine: (independent of growth factor support or transfusion within 7 days of study entry) neutrophils absolute value ≥1.5×109/L, platelets ≥75×109/L,
   2. Coagulation function：INR and APTT ≤2.5 times ULN，
   3. Blood biochemistry：total bilirubin ≤2 times ULN, AST or ALT≤2.5 times ULN;
   4. Renal function: Ccr ≥ 50 mL/min, total bilirubin, AST or ALT≤2.5 times ULN
7. Willing to take contraceptive measures during the trial period and within 3 months after the trial ends；
8. Voluntarily sign written informed consent before screening.

Exclusion Criteria:

1. Current or previous malignancy, unless radical therapy has been performed and there is no evidence of recurrence or metastasis in the past 5 years；
2. Patients scheduled for major surgery(examination for diagnostic purposes) within 4 weeks or participating in drug/device clinical trials;
3. Prior or concurrent indolent B-cell lymphoma transformation;
4. Have uncontrolled or significant cardiovascular disease, including:

   1. New York Heart Association (NYHA) Grade II or higher congestive heart failure, unstable angina, and myocardial infarction occurred within 6 months before the first administration of the study drug or arrhythmia needing treatment at the time of screening, LVEF <50%；
   2. Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmic right ventricular cardiomyopathy, restrictive cardiomyopathy, indeterminate cardiomyopathy)；
   3. Clinically significant QTc interval prolongation history, or QTc interval >470ms for female and >450ms for male in the screening period；
   4. Symptomatic coronary heart disease patients or needing treatment;
   5. Uncontrolled high blood pressure (on the basis of improving lifestyle, substandard blood pressure with reasonable and tolerable application of 2 or more antihypertensive drugs including diuretics for more than 1 month, or taking 4 or more antihypertensive drugs to control blood pressure effectively)；
5. Had active bleeding within 2 months prior to screening, or was taking anticoagulant drugs, or was considered by the investigator to have a clear tendency to bleeding;
6. Stroke or intracranial hemorrhage within 6 months；
7. Subjects with clinically significant gastrointestinal abnormalities that may affect drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
8. Active or uncontrolled HBV (HBsAg positive and HBV DNA titer positive), HCV Ab positive or HIV positive；
9. Uncontrolled, active systemic fungal, bacterial, viral, or other infections (defined as showing persistent signs/symptoms related to infection, despite the use of appropriate antibiotics or other treatments without improvement)；
10. Allergies or hypersensitivity reactions to orelabrutinib, rituximab or any other component of the applicable study drug;
11. Combined with drugs with moderate to severe inhibitory effect or strong induction effect on CYP3A;
12. Severe mental illness;
13. Expected survival <6 months
14. Pregnant and lactating women; For women of childbearing age who do not agree to use appropriate methods of contraception;
15. Poor compliance or inability to visit regularly;
16. Potentially life-threatening patients, or severe organ dysfunction, judged unsuitable for this trail by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | At the end of Cycle 6 (each cycle is 21 days)

SECONDARY OUTCOMES:
Occurrence of adverse events and serious adverse events | 3 years
  per cycle
progression-free survival (PFS) | 3 years
Overall survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, PhD, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China